CLINICAL TRIAL: NCT02498496
Title: MASTER-ED : Magnesium Sulfate to Prevent Hospitalisation of Acute Exacerbations of Chronic Obstructive Pulmonary Disease Seen in the Emergency Department
Brief Title: Magnesium Sulfate to Prevent Hospitalisation of Acute Exacerbations of Chronic Obstructive Pulmonary Disease
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: financing delays
Sponsor: Hôpital de Verdun (Other)
Responsible Party: Principal Investigator, Ivan Pavlov, Emergency Physician, Hôpital de Verdun
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MG-1
Record Dates: First submitted 2015-07-07; First posted 2015-07-15 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; AECOPD; Magnesium Sulfate; Acute exacerbation of COPD; Chronic Obstructive Pulmonary Disease; ED; ER; Emergency Department
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emergencies | interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnesium Sulfate (Experimental): Administration of a bolus dose of 2 g of MgSO4 in 100 mL of Normal Saline IV, in 20 min.
  Interventions: Drug: Magnesium Sulfate
- Placebo (Placebo Comparator): Administration of a bolus dose of 100 mL of Normal Saline, in 20 min.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Magnesium Sulfate — Administration of a bolus of 2 g of MgSO4 in 20 min, one dose.
  Other Names: Magnesium Sulfate Injection 50% Baxter. Number 5430
  Arms: Magnesium Sulfate
Drug: Placebo — Administration of 100 mL of Normal Saline
  Other Names: Normal saline 0.9 % Baxter 50 mL.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess whether administration of a bolus dose of MgSO4 (magnesium sulfate) plus standard therapy is superior to standard therapy alone for the management of Acute Exacerbations of Chronic Pulmonary Obstructive Disease (AECOPD) in the emergency department. The investigators hypothesize that MgSO4 causes faster recovery of the bronchospasm, and a reduction of the dead space, translating to the following clinical outcomes : less hospitalisation, lower length of stay (LOS), better composite outcome of hospitalisation + LOS + readmission for AECOPD.

DETAILED DESCRIPTION:
Patients presenting to the participant Emergency Departments (ED) with a diagnosis of AECOPD and who receive at least one dose of albuterol, will be randomized to receive either placebo or one dose of MgSO4 2g IV. Security and efficacy outcomes will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Current or previous smoking for at least 10 pack-years
* Confirmed COPD :

  1. reported by the patient if already diagnosed in the past by a pulmonary disease specialist or on the basis of respiratory function tests; or
  2. new diagnosis in the ED, with confirmatory pulmonary tests showing Forced Expiratory Volume (FEV1) / Forced Vital Capacity (FVC) ratio < 70% and FEV1< 80%
* Patient requires at least one dose of albuterol (salbutamol).

Exclusion Criteria:

* Dialysis patients
* Severe kidney disease, known or suspected to have a creatine clearance < 15.
* Metastatic neoplasm
* Patients who received IV MgSO4 in the last week.
* Hypotension, defined as systolic blood pressure less than 90.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2017-10 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of Admissions for AECOPD | baseline
  Number of patients admitted to hospital

SECONDARY OUTCOMES:
Recurrence of AECOPD | 10, 30, 90 days after hospital discharge
  A composite outcome of (death, re-admission for AECOPD, new visit for AECOPD in the ED) in patients who are discharged either directly from the ED or after admission on the wards.
Mortality of any cause | Participants will be followed for the duration of the hospital stay, an expected 2 weeks, and for 30 days after discharge, up to 1 year after randomization
Length of stay | Participants will be followed for the duration of the hospital stay, an expected 2 weeks, and up to 1 year after randomization.
  Measured in hours, from baseline to discharge, either from ED, or after hospital admission

OTHER OUTCOMES:
Respiratory failure requiring intubation | 72 hours after randomization
  Number of patients who require endotracheal intubation
Respiratory failure requiring non-invasive ventilation | 72 hours after randomization
  Number of patients who require non-invasive ventilation (CPAP, bilevel positive airway pressure (BiPAP) , Optiflow), excluding patients who were using non-invasive ventilation before baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Pavlov, MD, Principal Investigator — Hôpital de Verdun